CLINICAL TRIAL: NCT02026869
Title: Impact of Vaginal Administration of Metformin in Women With PCOS.
Brief Title: Vaginal Administration of Metformin in PCOS Patients.
Acronym: VMPCO
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, AHMED NASR, Professor, Assiut University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: Vaginal Metformin- Ahmed Nasr
Record Dates: First submitted 2014-01-02; First posted 2014-01-03 (Estimated); Last update posted 2014-01-03 (Estimated); Status verified 2014-01

CONDITIONS: PCOS
Keywords: Vaginal administration, PCOS, Metformin
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oral metformin (Active Comparator): Metformin 850 mg tablets taken by mouth every 12 hours for 6 months
  Interventions: Drug: Metformin
- Vaginal metformin (Active Comparator): Metformin 850 mg tablets taken vaginally every 12 hours for 6 months
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Metformin is taken either orally or vaginally every 12 hours
  Other Names: Cidophage

SUMMARY:
Polycystic ovary syndrome is a common cause of irregular periods, poor ovulation and delay in achieving pregnancy. Certain drugs may help improve ovarian activity in such women as metformin. Oral administration of metformin is accompanied by undesirable side effects. The vagina proved to be a good alternative to the oral route for other drugs. Using metformin through the vagina and avoidance of such side effects, while maintaining its effectiveness, would help women to better tolerate this drug.

DETAILED DESCRIPTION:
PCOS is the most common of all female endocrinopathies affecting 7-10% of women. A variety of drugs have been used to help improve follicular dynamics in PCOS patients. Metformin, an insulin sensitizer long known for its antidiabetic properties, has been used in PCOS patients. One of the major factors affecting compliance are the gastrointestinal side effects associated with oral administration of metformin. Knowing that the vagina is a good absorptive surface for many drugs, it is postulated that vaginal administration of metformin could be a good alternative to the oral route, if it proves effective. Both pharmacokinetic and clinical evidences of efficacy are traced for the vaginal route of administration.

ELIGIBILITY:
Inclusion Criteria:

* women with PCOS according to the Rotterdam criteria
* age 20-35 years
* not to have received any induction of ovulation in the preceding 3 months before enrollment

Exclusion Criteria:

* contraindications to metformin
* prior surgical management of PCOS

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2013-01; Primary Completion 2013-06 (Actual); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Ovulation rates | 6 months
  Ovulation rates assessed by transvaginal sonography (TVS) after oral versus vaginal administration of metformin in PCOS women.

SECONDARY OUTCOMES:
Therapeutic drug level | Over 24 hours after administration.
  Therapeutic drug levels are measured over 24 hours after oral and vaginal administration of metformin.

CONTACTS AND LOCATIONS:
Overall Officials: AHMED NASR, MD, Principal Investigator — Professor, Women's Health Hospital, Assiut University, Egypt.; MAGDY AMIN, MD, Study Director — Associate professor, dept. of Obstetrics & gynecology, Sohag University, Egypt
Locations (1):
- Women's Health Hospital, Asyut, Asyut Governorate, Egypt